CLINICAL TRIAL: NCT01265069
Title: Efficacy of 10-day Concomitant Regimen Versus High Dose Dual Therapy in Anti-Helicobacter Pylori Rescue Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201005064M
Record Dates: First submitted 2010-12-10; First posted 2010-12-22 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; concomitant therapy; high dose dual therapy; antibiotic resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high dose dual therapy (Active Comparator): Group A - high dose dual therapy (rabeprazole 20 mg qid, amoxicillin 750 mg qid for 14 days)
  Interventions: Drug: high dose dual therapy
- concomitant therapy (Experimental): Group B - concomitant therapy (rabeprazole 20 mg, amoxicillin 1000 mg, metronidazole 500 mg, clarithromycin 500 mg, bid for 10 days).
  Interventions: Drug: concomitant therapy

INTERVENTIONS:
Drug: high dose dual therapy — rabeprazole 20mg qid,amoxicillin 750mg qid for 14days
  Arms: high dose dual therapy
Drug: concomitant therapy — rabeprazole 20 mg,amoxicillin 1000 mg,metronidazole 500 mg,clarithromycin 500 mg, bid for 10 days
  Arms: concomitant therapy

SUMMARY:
Currently, a 10-day concomitant therapy has been reported to be equally effective and safe to the 10-day sequential therapy for 1st-line anti-Helicobacter pylori(H. pylori) therapy. To our knowledge, there has been no report concerning the efficacy of this regimen used as a rescue therapy.

The aims of this study are:

1. to compare the efficacy of high dose dual therapy and concomitant therapy as rescue regimen in H. pylori eradication;
2. to compare the patient adherence and adverse effects of these treatment regimens;
3. to investigate factors that may influence H. pylori eradication by these treatment regimens.

DETAILED DESCRIPTION:
Patients, aged 18, having H. pylori-positive chronic gastritis with/without peptic ulcers will be recruited. All undergo endoscopy with biopsy before treatment. Four to eight weeks after termination of treatment, H. pylori infection status will be examined by endoscopy with biopsy or the Carbon 13-urea breath test if the patients refuse the second endoscopy. The cytochrome P450 (CYP)2C19 genotype of each participant will be analyzed by the polymerase chain reaction-based restriction fragment length polymorphism (PCR-RFLP) method. A computed generated random numbers sequence will be blocked into two subgroups, say A and B.

If the patients had received anti-H. pylori therapy previously, they will be invited to enter the study for evaluating the efficacy of rescue regimens. After giving their written informed consent, all patients will be labeled with numbers by enrolling order. Each patient will be randomly allocated to one of two treatment groups which receives medications for 10 to 14 days:

group A - high dose dual therapy (rabeprazole 20 mg qid + amoxicillin 750 mg qid for 14 days); group B - concomitant therapy (rabeprazole 20 mg + amoxicillin 1000 mg + metronidazole 500 mg + clarithromycin 500 mg, bid for 10 days).

All patients will be asked to complete a questionnaire and to record symptoms and drug consumption daily in a diary card during the treatment period. Post-treatment, the patients will be seen at the Outpatient Clinic to investigate patient adherence and adverse effects of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients having H. pylori related chronic gastritis with/without peptic ulcers who are aged greater than 18 years and are willing to received eradication therapy.

Exclusion Criteria:

* pregnant or nursing woman
* serious concomitant illness and malignant tumor of any kind
* history of hypersensitivity to test drugs
* serious bleeding during the course of this ulcer
* previous gastric surgery
* receiving bismuth salts, proton pump inhibitors, or antibiotics in the previous month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
to compare the efficacy of 10-day concomitant regimen versus high dose dual therapy used as atni-Helicobacter pylori rescue therapy | 1.5 years
  The eradication rates (efficacy) will be evaluated by intention-to-treat (ITT) and per-protocol (PP) analysis.

SECONDARY OUTCOMES:
to compare the adverse effects and patient adherence of 10-day concomitant regimen versus high dose dual therapy used as atni-Helicobacter pylori rescue therapy | 1.5 years
  The safety and tolerability will be evaluated by the number of participant with adverse events and patient adherence (by counting unused medication after the treatment and record symptoms in a diary card).

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Chin Yang, M.D.Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan